CLINICAL TRIAL: NCT05935930
Title: Postoperative Effects of Propofol Versus Sevoflurane Anesthesia During Elective Non-Cardiac Surgeries. A Randomized Clinical Trial
Brief Title: Postoperative Effects of Propofol Versus Sevoflurane Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DTH: 22004
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-01

CONDITIONS: General Anesthetic Drug Adverse Reaction
Keywords: Cognitive function; General anesthesia; Inflammatory response; Oxidative stress; Propofol; Sevoflurane
MeSH Terms: interventions — Propofol; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (n=22) (Active Comparator): Propofol group
  Interventions: Drug: Propofol 10 MG/ML Injection
- Group S (n=22) (Active Comparator): Sevoflurane group
  Interventions: Drug: Sevoflurane Inhalation Liquid

INTERVENTIONS:
Drug: Propofol 10 MG/ML Injection — Propofol infusion
  Arms: Group P (n=22)
Drug: Sevoflurane Inhalation Liquid — Sevoflurane inhalation
  Arms: Group S (n=22)

SUMMARY:
Background: The choice of appropriate anesthetics is essential to protect brain function, decrease perioperative complications, and provide high-quality care, and better quality of life.

Objectives: To compare the efficacy and safety of propofol versus sevoflurane in patients undergoing elective, non-cardiac operations under general anesthesia.

Methods: This was a randomized (1:1), parallel, phase four clinical trial; carried out on 44 patients, who were candidates for elective, non-cardiac operations under general anesthesia at our hospital. Patients were randomly allocated into two equal groups in which anesthesia was maintained with propofol infusion in group P and sevoflurane inhalation in group S.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 years
* Body Mass Index (BMI) 25-35 kg/m2

Exclusion Criteria:

* ASA physical status > II
* Age < 21 years
* Patients with Montreal Objective Cognitive Assessment (MoCA-B) score < 24 points
* Patients with significant cardiovascular, cerebrovascular, respiratory, liver, renal, endocrine, blood, or immune diseases
* Patients with visual or auditory disease, infection, chronic inflammation, disturbance of consciousness, cognitive impairment, or dementia
* Patients on long-term use of sedatives or steroids, alcohol or drug abuse
* Allergy to any of the study drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Mean and Standard deviation of Neuron Specific Enolase enzyme (µg/L) in blood serum (mean±SD) | 24 hours after the end of operation
  Before operation (T0), 1 hour after the end of operation (T1), 24 hours the end of operation (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt